CLINICAL TRIAL: NCT04903847
Title: Changes in Weight After Switch to Dolutegravir/Lamivudine or Doravirine/Tenofovir/Lamivudine Compared to Continued Treatment With Dolutegravir/Tenofovir/Lamivudine for Virologically Suppressed HIV Infection. AVERTAS-2
Brief Title: Changes in Weight, Body Composition and Metabolic Parameters After Discontinuing Dolutegravir or Tenofovir Disproxil
Acronym: AVERTAS-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, MD, professor, dr.med., Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20012194
Record Dates: First submitted 2020-10-09; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Hiv; HIV Infections; HIV Lipodystrophy; Osteoporosis; Renal Insufficiency; Weight Gain; Obesity
Keywords: HIV; antiretroviral therapy; antiretroviral therapy adverse events; weight gain; body composition; fat distribution
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Osteoporosis; Renal Insufficiency; Weight Gain; Obesity | interventions — dolutegravir; Lamivudine; doravirine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Randomized controlled open-label superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dolutegravir/tenofovir disproxil/lamivudine (No Intervention): Continue dolutegravir 50 mg, tenofovir disproxil 245 mg, ,and lamivudine 300 mg once daily for 48 weeks.
- dolutegravir/lamivudine (Experimental): dolutegravir 50 mg/lamivudine 300 mg once daily for 48 weeks
  Interventions: Drug: Dolutegravir/Lamivudine 50 MG-300 MG Oral Tablet [DOVATO]
- doravirine/tenofovir disproxil/lamivudine (Experimental): 100 mg doravirin, 245 mg tenofovirdisoproxil and 300 mg lamivudine once daily for 48 weeks.
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100 MG-300 MG-300 MG Oral Tablet [DELSTRIGO]

INTERVENTIONS:
Drug: Dolutegravir/Lamivudine 50 MG-300 MG Oral Tablet [DOVATO] — Two-drug therapy
  Other Names: Dovato
  Arms: dolutegravir/lamivudine
Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100 MG-300 MG-300 MG Oral Tablet [DELSTRIGO] — Three-drug therapy
  Other Names: Delstrigo
  Arms: doravirine/tenofovir disproxil/lamivudine

SUMMARY:
Randomized controlled parallel open-label study in persons living with HIV. The aim is to study weight changes in patients switching from a dolutegravir and tenofovir disoproxil containing regimen to either a dolutegravir or tenofovir disoproxil free regimen.

DETAILED DESCRIPTION:
Randomized controlled parallel open-label study in persons living with HIV and at least 6 month of treatment with dolutegravir/abacavir/lamivudine prior to inclusion.

Participants (n=126) are randomized to continue 3 drug-regimen dolutegravir/tenofovir disoproxil/lamivudine (control) or switch to two-drug regimen with dolutegravir/lamivudine (intervention 1) or to three-drug regimen with doravirine/tenofovir disoproxil/lamivudine. Follow-up is 48 weeks. Data is collected at baseline and week 48.

Primary outcome is changes in weight from baseline of more than 2 kg.

Secondary outcomes are virus persistent viral suppression, changes in body composition and metabolism, changes in bone metabolisme and renal function, changes in liver elasticity and fat infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years old with diagnosed HIV and at least 6 months of ongoing treatment with dolutegravir/ doravirin/lamivudine will be included. Patients must have a plasma viral load (HIV-RNA) < 50 copies/ml at inclusion. For women of childbearing potential: Negative pregnancy test and willingness to use contraceptive (consistent with local regulations) during study period

Exclusion Criteria:

* Patients will be excluded in case of pre-existing viral resistance mutations to lamivudine, dolutegravir, tenofovir or doravirine the presence of hepatitis B antigen (HBsAg) or HBV DNA, cancer within past 5 years, pregnancy or breastfeeding. Any case of diabetes, cardiovascular disease or other chronic illness must be considered stable as assessed by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Body weight | 48 Weeks
  Primary outcome is a change in body weight of more than 2 kg from

SECONDARY OUTCOMES:
Virological control | 48 weeks
  Plasma HIV-RNA <50 copies/ml
Self-rated health | 48 weeks
  Changes in 12-item Short Form Health Survey (SF-12). Scores from 0 (worse) to 100 (best).
Insulin resistance | 48 weeks
  Impaired insulin resistance and/or β-cell function determined by changes in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Diabetic profile | 48 weeks
  Changes in HbA1c
Cholesterol profile | 48 weeks
  Changes in cholesterol total, HDL, LDL, VLDL
Fat distribution | 48 weeks
  Changes in Visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) determined by thoracic and upper abdominal CT-scan.
Hepatic elasticity | 48 weeks
  Changes in hepativ elasticity determined by liver elastography (Fibro-scan)
Hepatic fat infiltration | 48 weeks
  Changes in hepatic fat infiltration determined by liver elastography (Fibro-scan) and upper abdominal CT-scan
Body composition/perfiferal and central fat distribution | 48 weeks
  Changes in body fat distribtuion determined bu Dual Energy X-ray Absorbtiometry (DEXA)
Estimated Glomerular Filtration Rate (eGFR) (creatinine) | 48 weeks
  Changes in eGFR estimated by plasma creatinine
eGFR (cystatin) | 48 weeks
  Changes in estimated by plasma cystatin
Urea | 48 weeks
  Changes in plasma urea
Urine RBP/creatinine ratio | 48 weeks
  Changes in Urine RBP/creatinine ratio determined by spot urine Retinol Binding Protein (RBP) and creatinine analysis
Urine Beta-2-Microglobulin(B2M)/creatinine ratio | 48 weeks
  Changes in B2M/creatinine ratio determined by spot urine B2M and creatinine
Urine albumin/creatinine ratio | 48 weeks
  Changes in Urine albumin/creatinine ratio determined by spot urine albumine and creatinine analysis
Urine protein/creatinine ratio | 48 weeks
  Changes in urine protein/creatinine ratio determined by spot urine protein and creatinine analysis
Urine phosphate | 48 weeks
  Changes in spot urine phosphate
Bone mass density (BMD) | 48 weeks
  Changes in BMD assessed by DEXA
Bone-specific alkaline phosphate | 48 weeks
  Changes in plasma Bone-specific alkaline phosphate
Procollagen type 1 N-pro-peptide | 48 weeks
  Changes in procollagen type 1 N-pro-peptide
Type 1 collagen cross-linked C-telopeptide | 48 weeks
  Changes in plasma Type 1 collagen cross-linked C-telopeptide
Osteocalcin | 48 weeks
  Changes in plasma osteocalcin
Fasting ionized calcium | 48 weeks
  Changes in plasma fasting ionized calcium
25(OH)vitamin D vitamin D 25(OH)vitamin D | 48 weeks
  Changes in plasma 25(OH)vitamin D
Parathyroid hormone (PTH) vitamin D 25(OH)vitamin D | 48 weeks
  Changes in plasma parathyroid hormone (PTH)
Inflammation | 48 weeks
  High-sensitive C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Benfield, MD, Study Director — Center of Research and Disruption of Infectious Diseases
Locations (5):
- Denmark (5):
  - Department of Infectious Diseases, Aalborg University Hospital, Aalborg
  - Department of Infectious Diseases, Aarhus University Hospital, Aarhus
  - Department of Infectious Diseases, Rigshospitalet, Copenhagen
  - Department of Infectious Diseases, Hvidovre University Hospital, Hvidovre
  - Department of Infectious Diseases, Odense University Hospital, Odense

REFERENCES:
- [Background] Belloso WH, Orellana LC, Grinsztejn B, Madero JS, La Rosa A, Veloso VG, Sanchez J, Ismerio Moreira R, Crabtree-Ramirez B, Garcia Messina O, Lasala MB, Peinado J, Losso MH. Analysis of serious non-AIDS events among HIV-infected adults at Latin American sites. HIV Med. 2010 Oct 1;11(9):554-64. doi: 10.1111/j.1468-1293.2010.00824.x. Epub 2010 Mar 21. PMID 20345879
- [Background] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Background] Brown TT, Cole SR, Li X, Kingsley LA, Palella FJ, Riddler SA, Visscher BR, Margolick JB, Dobs AS. Antiretroviral therapy and the prevalence and incidence of diabetes mellitus in the multicenter AIDS cohort study. Arch Intern Med. 2005 May 23;165(10):1179-84. doi: 10.1001/archinte.165.10.1179. PMID 15911733
- [Background] Koethe JR, Jenkins CA, Lau B, Shepherd BE, Justice AC, Tate JP, Buchacz K, Napravnik S, Mayor AM, Horberg MA, Blashill AJ, Willig A, Wester CW, Silverberg MJ, Gill J, Thorne JE, Klein M, Eron JJ, Kitahata MM, Sterling TR, Moore RD; North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD). Rising Obesity Prevalence and Weight Gain Among Adults Starting Antiretroviral Therapy in the United States and Canada. AIDS Res Hum Retroviruses. 2016 Jan;32(1):50-8. doi: 10.1089/aid.2015.0147. Epub 2015 Sep 9. PMID 26352511
- [Background] Bakal DR, Coelho LE, Luz PM, Clark JL, De Boni RB, Cardoso SW, Veloso VG, Lake JE, Grinsztejn B. Obesity following ART initiation is common and influenced by both traditional and HIV-/ART-specific risk factors. J Antimicrob Chemother. 2018 Aug 1;73(8):2177-2185. doi: 10.1093/jac/dky145. PMID 29722811
- [Background] Hill A, Waters L, Pozniak A. Are new antiretroviral treatments increasing the risks of clinical obesity? J Virus Erad. 2019 Jan 1;5(1):41-43. doi: 10.1016/S2055-6640(20)30277-6. PMID 30800425
- [Background] Sax PE, Erlandson KM, Lake JE, Mccomsey GA, Orkin C, Esser S, Brown TT, Rockstroh JK, Wei X, Carter CC, Zhong L, Brainard DM, Melbourne K, Das M, Stellbrink HJ, Post FA, Waters L, Koethe JR. Weight Gain Following Initiation of Antiretroviral Therapy: Risk Factors in Randomized Comparative Clinical Trials. Clin Infect Dis. 2020 Sep 12;71(6):1379-1389. doi: 10.1093/cid/ciz999. PMID 31606734
- [Background] Burns JE, Stirrup OT, Dunn D, Runcie-Unger I, Milinkovic A, Candfield S, Lukha H, Severn A, Waters L, Edwards S, Gilson R, Pett SL. No overall change in the rate of weight gain after switching to an integrase-inhibitor in virologically suppressed adults with HIV. AIDS. 2020 Jan 1;34(1):109-114. doi: 10.1097/QAD.0000000000002379. PMID 31567162
- [Background] Vizcarra P, Vivancos MJ, Perez-Elias MJ, Moreno A, Casado JL. Weight gain in people living with HIV switched to dual therapy: changes in body fat mass. AIDS. 2020 Jan 1;34(1):155-157. doi: 10.1097/QAD.0000000000002421. PMID 31714355
- [Background] Nartey ET, Tetteh RA, Yankey BA, Mantel-Teeuwisse AK, Leufkens HGM, Dodoo ANO, Lartey M. Tenofovir-associated renal toxicity in a cohort of HIV infected patients in Ghana. BMC Res Notes. 2019 Jul 22;12(1):445. doi: 10.1186/s13104-019-4454-2. PMID 31331365
- [Background] Nishijima T, Kawasaki Y, Tanaka N, Mizushima D, Aoki T, Watanabe K, Kinai E, Honda H, Yazaki H, Tanuma J, Tsukada K, Teruya K, Kikuchi Y, Gatanaga H, Oka S. Long-term exposure to tenofovir continuously decrease renal function in HIV-1-infected patients with low body weight: results from 10 years of follow-up. AIDS. 2014 Aug 24;28(13):1903-10. doi: 10.1097/QAD.0000000000000347. PMID 25259702
- [Background] Casado JL, Santiuste C, Vazquez M, Banon S, Rosillo M, Gomez A, Perez-Elias MJ, Caballero C, Rey JM, Moreno S. Bone mineral density decline according to renal tubular dysfunction and phosphaturia in tenofovir-exposed HIV-infected patients. AIDS. 2016 Jun 1;30(9):1423-31. doi: 10.1097/QAD.0000000000001067. PMID 26919733
- [Background] Gupta SK, Yeh E, Kitch DW, Brown TT, Venuto CS, Morse GD, Ha B, Melbourne K, McComsey GA. Bone mineral density reductions after tenofovir disoproxil fumarate initiation and changes in phosphaturia: a secondary analysis of ACTG A5224s. J Antimicrob Chemother. 2017 Jul 1;72(7):2042-2048. doi: 10.1093/jac/dkx076. PMID 28369419
- [Background] Jacobson DL, Spiegelman D, Knox TK, Wilson IB. Evolution and predictors of change in total bone mineral density over time in HIV-infected men and women in the nutrition for healthy living study. J Acquir Immune Defic Syndr. 2008 Nov 1;49(3):298-308. doi: 10.1097/QAI.0b013e3181893e8e. PMID 18845956